CLINICAL TRIAL: NCT05782244
Title: Phase 2 Randomized Controlled Trial of Sildenafil Citrate for Treatment of Cerebrovascular Dysfunction in Chronic Traumatic Brain Injury
Brief Title: Sildenafil for Microvasculopathy in Chronic TBI
Acronym: CVR-TBI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 852199
Record Dates: First submitted 2022-11-22; First posted 2023-03-23 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Sildenafil citrate low dose (Active Comparator): Sildenafil citrate 20 mg, oral, TID
  Interventions: Drug: Sildenafil Citrate low dose
- Placebo (Placebo Comparator): Placebo, oral, TID
  Interventions: Drug: Placebo
- Sildenafil citrate medium dose (Active Comparator): Sildenafil citrate 40 mg, oral, TID
  Interventions: Drug: Sildenafil medium dose
- Sildenafil citrate high dose (Active Comparator): Sildenafil citrate 80 mg, oral, TID
  Interventions: Drug: Sildenafil high dose

INTERVENTIONS:
Drug: Sildenafil Citrate low dose — Sildenafil citrate 20 mg, oral, TID
  Other Names: Sildenafil lowest dose
  Arms: Sildenafil citrate low dose
Drug: Placebo — Placebo, oral, TID
  Other Names: Masked placebo
  Arms: Placebo
Drug: Sildenafil medium dose — Sildenafil 40 mg, oral, TID
  Other Names: Sildenafil middle dose
  Arms: Sildenafil citrate medium dose
Drug: Sildenafil high dose — Sildenafil 80 mg, oral, TID
  Other Names: Sildenafil highest dose
  Arms: Sildenafil citrate high dose

SUMMARY:
Traumatic Cerebral Vascular Injury (TCVI) is a common consequence of traumatic brain injury (TBI), including mild TBI (mTBI). TCVI is associated with poor recovery after TBI in animal models. TCVI can be measured non-invasively in humans, and therapies targeting TCVI are attractive candidates to ameliorate the consequences of TBI. Sildenafil potentiates nitric oxide (NO) dependent vasodilatation and is approved by the Food and Drug Administration (FDA) for the treatment of erectile dysfunction and primary pulmonary hypertension. In pre-clinical models of stroke, sildenafil improves cerebral blood flow (CBF), promotes, angiogenesis, neurogenesis and improves recovery. In an initial Phase 2a trial (NCT01762475) of sildenafil in patients with chronic moderate to severe TBI, the investigators found that low dose sildenafil (25 mg BID) therapy is safe and well tolerated, that a single dose of sildenafil 50 mg potentiates CVR in areas of the brain with dysfunctional endothelium, and that CVR is a reliable diagnostic marker of TCVI and has potential as a pharmacodynamic and predictive biomarker. In this proposal, the investigators will conduct a randomized clinical trial to determine the optimal PDE5 inhibitor dose to improve or normalize microvascular function (as measured by the change in CVR measurements before and after a single dose of sildenafil, or ΔCVR) using a range of sildenafil citrate doses: 20, 40, 80 mg) in chronic TBI patients. The investigators will also test the safety and tolerability of the same dose ranges of chronic (4-week) thrice daily sildenafil or placebo administration in chronic TBI patients and explore its effects on chronic symptoms and clinical outcomes.

DETAILED DESCRIPTION:
Objectives:

Objective 1: To determine the optimal sildenafil dose to improve microvascular function (ΔCVR measure) after a single dose (dose range sildenafil 20-80 mg) in 160 chronic TBI patients.

Objective 2: To assess the safety and tolerability of a range of PDE5 inhibitor doses (placebo, sildenafil 20, 40, 80 mg, administered orally three times daily (TID)) in 160 chronic TBI subjects.

Objective 3 (exploratory): To measure the effect of chronic (4-week) PDE-5 inhibitor administration at 3 different doses compared to placebo on TBI symptom self-report, clinician-administered outcome measures, and clinician interview-based impression of change.

Primary Endpoint: The primary outcome measure will be the baseline visit delta cerebrovascular reactivity (ΔCVR) or the difference between global CVR (mm/Hg) measured before and 1 hour after a randomized, double blind, oral administration of one of 3 doses of sildenafil (20mg, 40 mg or 80 mg) or placebo. CVR (mm/Hg) is an imaging measure of cerebral microvascular function and is measured in the MRI nd by the change in the fMRI-BOLD signal during a 7 minute 5% hypercapnia challenge (alternating inhalation of room air and room air enriched with 5% CO2 in a block design for 1 minute each over 7 minutes total).

Secondary Endpoints: The secondary outcome measures will be an assessment of study drug safety and tolerability. Safety will be measured by the number of participants with treatment-related adverse events as assessed by the CTCAE v4.0. Tolerability will be measured the number of participants with treatment-related adverse events as assessed by the CTCAE v4.0, self-report compliance with drug regimen and remaining pill count at the end of the study.

Exploratory Endpoints: Clinician administered and self-report measures of clinical symptom improvement, change in neurocognitive function and post-concussive symptoms improvement before and after 4 week sildenafil intervention. These will be measured by the change in baseline and end of treatment testing/reports of the following functional and symptom neurobehavioral measures: Clinician Interview-Based Impression (CIBI); Glasgow Outcome Scale-Extended (GOSE); Rivermead Post-Concussion Symptom Questionnaire (RPQ); Headache Impact Test-6 (HIT-6); PTSD Checklist for DSM-5- Civilian Version (PCL-5); Patient Health Questionnaire 9 (PHQ-9); Mental Fatigue Scale (MSF); NeuroQOL Short form for Positive Affect and Well Being; NeuroQOL Short form for Cognitive Functioning in Everyday Activities; Rey Auditory Verbal Learning Test (RAVLT); Brief Visuospatial Memory Test-Revised (BVMT-R); Trail Making Tests A and B (TMT); Processing Speed Index (PSI); Digit Symbol and Symbol Search of the Wechsler Adult Intelligence Scale (WAIS-IV); Simple and Complex Visual Reaction Time; Delis Kaplan Verbal Fluency Test (DKVFT); Grooved Pegboard Test; Brief Test of Adult Cognition by Telephone (BTACT).

Study Population: The study population for this protocol consists of 160 chronic TBI patients between the ages of 18 and 55 (both men and women) who have suffered a TBI more than 6 months before enrollment and remain symptomatic with at least 3 persistent post-concussive symptoms. The patients will be recruited from the University of Pennsylvania Health System (UPenn) and the Walter Reed National Military Medical Center (WRNMMC) TBI clinics and clinic referrals.

Phase: II

Description of Sites/Facilities : This is a two-site study, conducted at Penn Presbyterian Medical Center (PPMC), the Level I Trauma Center for UPenn, and WRNMMC, the flagship hospital for the Military Health System. Both PPMC and WRNMMC are major referral centers for TBI. The Clinical TBI Center at PPMC, led by Dr. Diaz-Arrastia, evaluates over 200 acute TBI cases admitted to the hospital per year and maintains an active outpatient TBI clinic that annually evaluates and treats over 800 unique TBI patients. WRNMMC is a tertiary referral center for active duty military personnel medically evacuated for TBI and has a specialized outpatient center for the evaluation and treatment of chronic TBI, the National Intrepid Center of Excellence (NICoE), which annually evaluates and treats 300-400 chronic TBI patients.

Enrolling Sites: Two (University of Pennsylvania Health System, Philadelphia, PA and Walter Reed National Military Medical Center, Bethesda, MD)

Description of Study Intervention: Sildenafil citrate is a phosphodiesterase-5 (PDE-5) inhibitor that is FDA-approved and widely used as a therapy for primary pulmonary hypertension and erectile dysfunction. Sildenafil or placebo will be administered at 3 doses (20mg, 40mg, 80mg) to the study participants to assess both single dose effect on CVR as well as safety, tolerability, and (as an exploratory measure) efficacy after 4-week thrice daily oral administration.

Study Duration: 48 months (i.e., 4 years)

Participant Duration:1 month

ELIGIBILITY:
Inclusion Criteria

To be eligible to participate in this study, an individual must meet all of the following criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged 18-70
4. Defense Enrollment Eligibility Reporting System (DEERS) eligible (WRNMMC only; N/A for UPenn)
5. History of TBI greater than 6 months and less than 25 years prior to enrollment, based on the 2023 American Congress of Rehabilitation Medicine Criteria92;

   1. Plausible Mechanism of Injury: Criterion 1 focuses on the external force that likely disrupted brain function, including blast/explosion forces and acknowledging intentional causes.
   2. Clinical Signs: Criterion 2 highlights signs observed or elicited during examination, distinguishing them from subjective symptoms.
   3. Acute Symptoms: Criterion 3 considers subjective acute symptoms, requiring at least two symptoms to be present.
   4. Clinical Examination/Laboratory Findings: Criterion 4 is a new addition, incorporating findings like cognitive impairment or oculomotor impairment.
   5. Neuroimaging: While not required for diagnosis, neuroimaging can be used to provide further evidence of brain injury.
6. Chronic persistent post-concussive symptoms (Symptom Score > 1 on at least 3 items from the Rivermead Post-Concussion Symptom Questionnaire; RPQ)
7. Glasgow Outcome Scale-Extended (GOSE) between 5-7
8. Ability to take oral medication and be willing to adhere to the study intervention regimen
9. Ability to participate in and complete 1 MRI including 2 CVR challenges and 4-week treatment period.
10. Adequate hearing and vision based on self-report and examiner's observation

Exclusion Criteria

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Contraindication to sildenafil which includes the following:

   1. Current/ongoing (within past month) use of organic nitrate vasodilators or riociguat
   2. Current/ongoing (within past month) use of ritonavir (HIV-protease inhibitor)
   3. Current/ongoing (within past month) use of erythromycin, ketoconazole, or itraconazole
   4. Current/ongoing (within past month) use of cimetidine
   5. Current resting hypotension (BP < 90/50 mm Hg)
   6. Current severe renal insufficiency
   7. Current hepatic cirrhosis
   8. Current cardiac failure or coronary artery disease causing unstable angina
   9. Retinitis pigmentosa
   10. Known hypersensitivity or allergy to sildenafil of any of its components
   11. History of melanoma or suspicious skin lesions for melanoma on skin examination
2. Daily therapy with a PDE5 inhibitor within the month prior to consent
3. History of penetrating TBI
4. History of disabling neurological or psychiatric disorder not related to TBI
5. Active substance abuse or dependence during the past 6 months
6. Estimated preinjury intellectual level ≤70 (based on educational and vocational history)
7. Inability to understand written and spoken English, in the opinion of the investigator
8. Current inclusion in another interventional trial
9. Subjects with metal implants that would interfere with the MR imaging procedures
10. History of priapism
11. Pregnant or breast-feeding women
12. Actively suicidal (based on clinician assessment OR if patient endorses item 9 on Patient Health Questionnaire 9 (PHQ-9) and endorses suicidal ideation on Columbia Suicide Severity Rating Scale(CSSRS)
13. Hypertension requiring treatment with more than two antihypertensive drugs
14. Hyperlipidemia requiring treatment with more than one lipid lowering drug
15. Diabetes mellitus requiring medical treatment with insulin

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-07-02 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Optimal Dose | Assessed at baseline visit
  Delta cerebrovascular reactivity (ΔCVR) after single-dose sildenafil administration during the neuroimaging session.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Assessed over 4 week daily intervention of 3 doses of sildenafil in TBI patients
  Safety will be measured by the number of participants with treatment-related adverse events as assessed by the CTCAE v4.0. Tolerability will be measured the number of participants with treatment-related adverse events as assessed by the CTCAEv4.0, and by number of participants who did not complete the course of treatment. Compliance will be measured by self-report compliance with drug regimen and pill counts remaining at the end of the study.

OTHER OUTCOMES:
Clinician Interview-Based Impression (CIBI) | Assessed at baseline and at the end of the 4 week intervention.
  Change in clinical status, neurocognitive function and post-concussive symptoms between baseline and completion of a 4 week sildenafil intervention, measured by the change in baseline and end of treatment using the Clinician Interview-Based Impression (CIBI) measure.
Glasgow Outcome Scale-Extended (GOSE) | Assessed at baseline and at the end of the 4 week intervention.
  Change in clinical status, neurocognitive function and post-concussive symptoms between baseline and completion of a 4 week sildenafil intervention, measured by the change in baseline and end of treatment using the Glasgow Outcome Scale-Extended (GOSE) measure.

CONTACTS AND LOCATIONS:
Overall Officials: Ramon Diaz-Arrastia, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Kalyani P, Lippa SM, Werner JK, Amyot F, Moore CB, Kenney K, Diaz-Arrastia R. Phosphodiesterase-5 (PDE-5) Inhibitors as Therapy for Cerebrovascular Dysfunction in Chronic Traumatic Brain Injury. Neurotherapeutics. 2023 Oct;20(6):1629-1640. doi: 10.1007/s13311-023-01430-z. Epub 2023 Sep 11. PMID 37697134